CLINICAL TRIAL: NCT00212836
Title: A Multicenter, Double-Blind, Flexible -Dose, 6-Month Trial Comparing the Efficacy Safety of Asenapine With Olanzapine in Stable Subjects With Predominant, Persistent Negative Symptoms of Schizophrenia
Brief Title: Efficacy and Safety of Asenapine Compared With Olanzapine in Patients With Persistent Negative Symptoms of Schizophrenia (25543)(COMPLETED)(P05817)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05817; Aphrodite;; 25543
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — asenapine; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine (Experimental)
  Interventions: Drug: asenapine
- Olanzapine (Active Comparator)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: asenapine — 5-10 mg sublingually twice daily for 26 weeks
  Arms: Asenapine
Drug: olanzapine — 5-20 mg by mouth once daily for 26 weeks
  Other Names: Zyprexa
  Arms: Olanzapine

SUMMARY:
Treatment with conventional antipsychotics such as haloperidol has little effect or may sometimes even worsen negative symptoms (such as blunted affect, emotional withdrawal, and poor rapport) of schizophrenia. The newer "atypical" antipsychotics agents, such as olanzapine, have shown improvement in the treatment of negative symptoms in acute trials. The purpose of this study is to compare an investigational compound (asenapine) with a marketed agent (olanzapine) in the treatment of stable subjects with persistent negative symptoms of schizophrenia for 6 months. Patients completing this study may be eligible to participate in an extension 6 months of treatment. Patients are required to have stable symptoms prior to entry into study.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented current diagnosis of schizophrenia of paranoid, disorganized, catatonic, residual, or undifferentiated subtype with persistent negative symptoms.
* No increase in level of psychiatric care during the past few months due to worsening of symptoms of schizophrenia.
* Caregiver required.

Exclusion Criteria:

* Have an uncontrolled, unstable clinically significant medical condition.
* Have any other psychiatric disorder other than schizophrenia as a primary diagnosis including depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2005-04-21 (Actual); Primary Completion 2007-06-15 (Actual); Study Completion 2007-08-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline at 6-months in Negative symptoms of schizophrenia measured by the Negative Symptoms Assessment (NSA) scale | Change from baseline at 6-months

SECONDARY OUTCOMES:
Change from baseline at 6-months in quality of life measured by the Quality of Life (QLS) scale | Change from baseline at 6-months
Positive and negative symptoms and other symptoms of schizophrenia e.g., hostility, excitement, disorganized thoughts and cognition measured by the Positive and Negative Symptom Scale (PANSS) | Change from baseline at 6-months
Depressive symptoms measured by the Calgary Depression Scale for Schizophrenia (CDSS) | Change from baseline at 6-months
Overall clinical global impression of severity improvement measured by the Clinical Global Impression of Severity (CGI-S) and Clinical Global Impression of Improvement (CGI-I) | Change from baseline at 6-months

REFERENCES:
- [Result] Buchanan RW, Panagides J, Zhao J, Phiri P, den Hollander W, Ha X, Kouassi A, Alphs L, Schooler N, Szegedi A, Cazorla P. Asenapine versus olanzapine in people with persistent negative symptoms of schizophrenia. J Clin Psychopharmacol. 2012 Feb;32(1):36-45. doi: 10.1097/JCP.0b013e31823f880a. PMID 22198451